CLINICAL TRIAL: NCT05895942
Title: Exploring the Molecular Mechanism of Secondary Resistance to Imatinib in Gastrointestinal Stromal Tumors Based on KIT Mutation
Brief Title: Exploring the Molecular Mechanism Based on KIT Mutation
Acronym: EMMBKM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TQXB-GIST-001
Record Dates: First submitted 2022-07-19; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2022-07

CONDITIONS: GIST
MeSH Terms: interventions — Imatinib Mesylate; Coal Tar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — stool specimen Serum Specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Imatinib treatment group: Chinese patients with unresectable C-kit9/11-mutated GIST were selected as the research subjects, and the therapeutic effect was observed after standard treatment with imatinib mesylate
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — The control group, before and after imatinib treatment, and patients with different efficacy of imatinib treatment were collected, and the correlation analysis was performed to screen the key flora and metabolites that affect the efficacy of imatinib
  Other Names: treat

SUMMARY:
Imatinib remains suboptimal for recurrence/metastasis and unresectable GIST response rates. With the maturity of genomics and metabolomics, people gradually realize the role of gut microbiota in tumor therapy. The gut microbiota may affect tumor treatment by regulating the tumor microenvironment or the host immune system, and some bacteria can fight tumors by activating the immune system. Growing evidence shows that the effect of tumor therapy is related to the composition of the gut microbiota of patients, and that the composition of the gut microbiota of patients sensitive to drug treatment has certain characteristics, and these characteristics may be used as biomarkers to predict the prognosis of treatment. At present, it remains unclear whether the efficacy of imatinib is related to the gut microbiota in GIST patients. Therefore, precise mining of microbial information and the development of reasonable and feasible microbial interventions are expected to optimize the treatment strategy of GIST to a large extent and provide a basis for individualized treatment of advanced GIST.

DETAILED DESCRIPTION:
Taking Chinese patients with unresectable C-kit9/11-mutated GIST as the research object, the treatment effect was observed after standardized treatment with imatinib mesylate. To explore the relationship between intestinal flora and the efficacy of imatinib treatment, to find new biomarkers to predict the efficacy of imatinib, and to provide reference for individualized treatment of imatinib

ELIGIBILITY:
Inclusion Criteria:

* BMI index 18.5-23.9kg/m2;
* Pathologically diagnosed patients with unresectable GIST, and genetic testing is C-kit9/11 mutation;
* No previous surgery;
* ECOG score: 0-1 points;
* Expected survival period ≥ 6 months;
* All patients should have measurable or evaluable target lesions;
* Able to eat liquid diet The above; no complete gastrointestinal obstruction or perforation; no distant metastasis;
* The main organ functions are normal, that is, the following criteria are met:

  1. The blood routine examination standards must be met (no blood transfusion and blood products within 14 days, no G-CSF use) and other hematopoietic stimulating factors): a) HB≥80 g/L; b) ANC≥1.5×109/L; c) PLT≥100×109/L;
  2. Biochemical tests should meet the following criteria: a) TBIL <1.5×ULN; b) ALT and AST<2.0×ULN; c) Serum Cr≤1.5×ULN or endogenous creatinine clearance rate> 50 mL/min (Cockcroft-Gault formula);
  3. Pulmonary function assessment of normal lung function or mild to moderate abnormality (VC%>60%, FEV1>1.2L, FEV1%>40%, DLco>40%);
  4. Cardiovascular function evaluation: cardiac function grades I to II;
* Have certain self-care Ability and language comprehension.

Exclusion Criteria:

* 1. Patients with pathological types and primary tumor sites that do not meet the inclusion criteria;
* 2. There is a risk of gastrointestinal perforation;
* 3. Has undergone surgical treatment;
* 4. Have ever suffered from malignant tumor;
* 5. Those with a history of severe lung or heart disease;
* 6. Active infection or unexplained fever >38.5℃ within 2 weeks before randomization;
* 7. Known major active infection, or the investigator judges that there is a major blood, renal, metabolic, gastrointestinal or endocrine dysfunction;
* 8. Those with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* 9. The subject has active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method);
* 10. Those who have been vaccinated with live vaccines within 3 months before treatment;
* 11. During acute or chronic tuberculosis infection (positive T-spot test and suspected tuberculosis foci on chest X-ray);
* 12. Those with a history of drug, drug or alcohol abuse (drinking ≥5 times a week, etc.);
* 13. Intravenous infusion cannot be performed;
* 14. Severe diarrhea in the past 2 months (watery stools ≥ 3 times per day and lasted ≥ 3 days);
* 15. Severe constipation (≤2 times of defecation per week with difficulty in defecation) in the past 2 months;
* 16. Antibiotics have been used in the past 2 months for 3 days or more;
* 17. Have used proton pump gastric drugs, acid suppressants, mucosal protective agents, opioid psychotropic drugs, hormones, immunosuppressants, cytotoxic drugs and other drugs within the past 2 months for 3 days or more;
* 18. Have used probiotics, prebiotics or synbiotic within the past 2 months for 3 days or more;
* 19. Received drug treatment for the following diseases in the past 1 month: cholecystitis, peptic ulcer, urinary tract infection, acute pyelonephritis, cystitis, hyperthyroidism and other abnormal thyroid function;
* 20. Gastrointestinal surgery, appendicitis surgery, enema, colon cleansing and other medical operations within the past 1 year;
* 21. During pregnancy and lactation (women) or lactose intolerance;
* 22. Patients with high blood pressure that cannot be reduced to the normal range after antihypertensive drug treatment (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg); patients with a history of unstable angina pectoris; newly diagnosed within 3 months before screening Angina pectoris or myocardial infarction within 6 months before screening; arrhythmia (including QTcF: ≥450 ms for men, ≥470 ms for women) requires long-term use of antiarrhythmic drugs and New York Heart Association classification ≥ grade II cardiac insufficiency;
* 23. According to the judgment of the investigator, the subject has other factors that may cause him to be forced to terminate the study halfway, such as suffering from other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory test values, family or social factors, Situations that may affect the safety of subjects or the collection of trial data;
* 24. The investigator judges other circumstances that may affect the conduct of clinical research and the judgment of research results;
* 25. Research center staff, researcher's partner or first-degree relative;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese patients with unresectable C-kit9/11-mutated GIST
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Degree of tumor regression | 6 months
  We used the RECIST 1.1 evaluation criteria to evaluate the response to the imatinib therapy and accordingly divided patients into two groups,Response and No Response.

CONTACTS AND LOCATIONS:
Overall Officials: jun j Yang, Master, Study Chair — The First Affiliated Hospital of Air Force Medicial University
Locations (1):
- Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No